CLINICAL TRIAL: NCT04827706
Title: Occurrence, Trends, Management and Outcomes of Patients Hospitalized With Myocarditis - Ten-year Perspectives From the MYO-PL Nationwide Database
Brief Title: Occurrence, Trends, Management and Outcomes of Patients Hospitalized With Myocarditis
Acronym: MYO-PL
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Other Study IDs: MYO-PL
Record Dates: First submitted 2021-03-08; First posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Myocarditis; Sudden Cardiac Death; Cardiomyopathies; Arrythmia; Heart Failure
Keywords: cardiomyopathy; children; endomyocardial biopsy; epidemiology; heart failure; cardiac magnetic resonance
MeSH Terms: conditions — Myocarditis; Death, Sudden, Cardiac; Cardiomyopathies; Arrhythmias, Cardiac; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The epidemiology of myocarditis is largely unknown and based mainly on small single-center studies. The study aim to evaluate the current incidence, clinical characteristics and outcomes of patients hospitalized due to myocarditis in a general population.

DETAILED DESCRIPTION:
In this retrospective-prospective study, data from the National Health Fund (NHF), which is the only public healthcare insurer in Poland is used. The NHF reimburses drugs and healthcare services provided by healthcare providers (both public and private) with public funds collected from health insurance premiums. In Poland, public health insurance is obligatory for almost all Poles - in December 2019, 88.4% of approx. 38 million Poles had public health insurance and were entitled to obtain healthcare services and drugs reimbursed by the NHF.

Based on NHF claims data, the healthcare services reported over the years 2009-2021 with a diagnosis of myocarditis - hospitalizations reported with codes I40, I40.0, I40.1, I40.8, I40.9, I41, I41.0, I41.1, I41.2, I41.8, I51.4, B33.2 are derived according to the International Classification of Diseases and Related Health Problems, 10th Revision (ICD-10). The dataset is narrowed to the first myocarditis hospitalization, i.e. patients for whom no information about the diagnosis of myocarditis is reported in the 400 days preceding the hospitalization. For such a group of patients, and to establish the baseline characteristics of the patients, data is analyzed 400 days back from the initial diagnosis of myocarditis. Also, in-hospital and long-term outcomes are analyzed, including all-cause mortality as well as the occurrence of selected diseases (defined as receiving a service where selected ICD-10 was reported), and selected procedures are obtained, defined with codes according to International Classification of Diseases, 9th Revision, Clinical Modification (ICD-9-CM). For the follow-up, at least a six-month period is required.

To show differences related to the age of patients hospitalized due to myocarditis, baseline characteristics and long-term outcomes are assessed with regard to age groups.

Data from the Central Statistical Office of Poland is also used to refer the obtained results to the population of Poland and to obtain life tables for survival analysis.

No specific exclusion criteria were applied. No ethics approval was required for this study, as it involved the analysis of administrative data.

ELIGIBILITY:
Inclusion Criteria:

* first myocarditis hospitalization

Exclusion Criteria:

* no specific exclusion criteria were applied

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with first myocarditis hospitalization in Poland in observed time period.
Sampling Method: Probability Sample
Enrollment: 19978 (Actual)
Dates: Start 2009-01-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Characteristics of myocarditis in Poland | 10 years
  Distribution of myocarditis incidence regarding to voivodeship/ district, city size (number of residents), hospital and ward type of admission
Seasonal occurrence | 10 years
  Seasonal occurrence rate of myocarditis regarding to gender and age
In-hospital mortality | 10 years
  Occurrence of all-cause death during initial hospitalization for myocarditis
Long-term mortality | 10 years
  Occurrence of all-cause death at 10-year observation.
Analysis of in-hospital course of patients with myocarditis. | 10 years
  Hospitalization length
Trends in the utilisation rate of diagnostic procedures. | 10 years
  Trends in the application rate of diagnostic procedures aimed at diagnosing myocarditis (i.e. cardiac magnetic resonance, endomyocardial biopsy, troponin, echocardiography, coronary angiography)
Occurrence of recurrent myocarditis | 10 years
  Occurrence of recurrent hospitalization for myocarditis
Occurrence of heart failure | 10 years
  Occurrence of heart failure hospitalization after diagnosis of myocarditis

CONTACTS AND LOCATIONS:
Overall Officials: Marcin Grabowski, Professor, Study Chair — Medical University of Warsaw; Grzegorz Opolski, Professor, Study Chair — Medical University of Warsaw
Locations (1):
- First Department of Cardiology, Medical University of Warsaw, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Undecided
data can be provided upon request

REFERENCES:
- [Derived] Ozieranski K, Tyminska A, Chabior A, Kruk M, Kon B, Maciejewski C, Opolski G, Grabowski M. Sex differences in incidence, management, and outcomes in adult patients aged over 20 years with clinically diagnosed myocarditis in the last 10 years: data from the MYO-PL nationwide database. Pol Arch Intern Med. 2022 Apr 28;132(4):16199. doi: 10.20452/pamw.16199. Epub 2022 Jan 27. PMID 35084153
- [Derived] Ozieranski K, Tyminska A, Kruk M, Kon B, Skwarek A, Opolski G, Grabowski M. Occurrence, Trends, Management and Outcomes of Patients Hospitalized with Clinically Suspected Myocarditis-Ten-Year Perspectives from the MYO-PL Nationwide Database. J Clin Med. 2021 Oct 12;10(20):4672. doi: 10.3390/jcm10204672. PMID 34682794